CLINICAL TRIAL: NCT05940181
Title: A Safety and Efficacy Study of XH001 (Neoantigen Cancer Vaccine) Combined With Sintilimab Injection in Advanced Solid Tumors
Brief Title: A Safety and Efficacy Study of XH001 Combined With Sintilimab Injection in Advanced Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: jianming xu (Other)
Collaborators: NeoCura (Industry)
Responsible Party: Sponsor-Investigator, jianming xu, Director, Head of Department of Oncology, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Organization: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XKY-C-001
Record Dates: First submitted 2023-05-11; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumor
Keywords: cancer vaccine; mRNA; neoantigen

STUDY DESIGN:
Intervention Model Description: single-center, open-label, single-arm, dose escalation exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XH001+ sintilimab (Experimental): XH001: 2 dose level Sintilimab: 200mg iv, 21 day per cycle
  Interventions: Biological: XH001+ sintilimab

INTERVENTIONS:
Biological: XH001+ sintilimab — During treatment period, subjects will receive 6 cycles of XH001+ sintilimab, followed by sintilimab monotherapy (sintilimab will be administered for up to 18 cycles or for 1 year, whichever comes first).

SUMMARY:
This is an investigator-initiated, single-center, open label, single-arm dose escalation study of XH001 (neoantigen tumor vaccine) in combination with sintilimab for advanced solid tumors. To evaluate the safety and tolerability of XH001 combined with sintilimab in subjects with advanced solid tumors, and preliminarily evaluate the efficacy of the combination therapy in subjects with advanced solid tumors.

The study will include pre-screening period (about 12 weeks), screening period (Weeks -4 to Day 1, and Week -1 to Day -1 will be baseline period), treatment period (Day 1 to Week 16 will be combination treatment period, followed by sintilimab monotherapy), and follow-up period. After signing pre-screening informed consent, tumor tissue and blood samples will be collected for gene sequencing, neoantigen prediction and vaccine preparation. During vaccine preparation, subjects will receive sintilimab (200mg, intravenous infusion, 21-day per cycle) or other antitumor therapy as deemed appropriate by the investigator. Subjects who sign and provide formal informed consent will enter the formal screening period, and qualified subjects will enter treatment period. During the treatment period, subjects will receive 6 cycles of XH001+ sintilimab, followed by sintilimab monotherapy (sintilimab will be administered for up to 18 cycles or for 1 year, whichever comes first).

The dose escalation phase follows standard 3+3 design. 9-12 subjects are expected to be enrolled at 2 given dose level.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial.
* Is ≥18 years and ≤ 75 years of age on day of signing informed consent.
* Has a histologically confirmed advanced solid tumor. Subjects must have documented progression after standard therapy or is intolerant of, refuses, or is not eligible for standard therapy.
* Has at least 1 measurable disease lesion as defined by Response Evaluation Criteria in Solid Tumors.
* Has a life expectancy of ≥12 weeks.
* Has an ECOG performance status of 0-1.
* Has adequate organ function as confirmed by laboratory values listed in the main body of the protocol

Exclusion Criteria:

* Subject who need to receive systemic application of anti-allergic drugs for a long time, or have a history of life-threatening allergic reactions to any vaccine or drug;
* Symptomatic or rapidly progressive central nervous system metastases. Patients with extensive lung metastases resulting in dyspnea; patients with tumors close to or invading major blood vessels or nerves;
* New cerebrovascular accident (including ischemic stroke, hemorrhagic stroke, and transient ischemic attack) within 6 months before screening;
* Subject with acute myocardial infarction within 6 months before screening, or uncontrolled angina, uncontrolled arrhythmia, severe heart failure (see Appendix 3, New York Heart Association Heart Failure Classification Criteria NYHA Class ≥ III) and other cardiovascular diseases;
* Subject who have received treatment with immunomodulatory drugs 4 times before the first vaccination day (D1), including but not limited to: IL-2, CTLA-4 inhibitors, CD40 agonists, CD137 agonists, IFN-α (except for high-risk surgical subjects who use IFN-α as adjuvant therapy, if IFN-α treatment is stopped 4 times before this trial);
* Subject who received blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) before baseline;
* Subject with skin diseases (e.g., psoriasis) at baseline that may prevent the intradermal injection of vaccine into the target area;
* Subject still suffer from adverse reactions (except alopecia and platinum-induced neurotoxicity ≤ grade 2) that have not been restored to CTCAE version 5.0 grade ≤ 1 after previous anti-tumor treatment during the screening period;
* Concomitant use of steroid hormone drugs (tumor or non-tumor related diseases) is required; however, topical application (not applied to the vaccination site) or inhaled steroid drugs are required;
* Subject has an active infection or uncontrollable infection (except for simple urinary tract infection or upper respiratory tract infection) requiring systemic treatment;
* Subjects with positive human immunodeficiency virus antibody, hepatitis B surface antigen and/or hepatitis B core antibody and positive hepatitis B virus deoxyribonucleic acid > 1000 IU/mL, hepatitis C virus antibody, Treponema pallidum-specific antibody in virological monitoring during the screening period;
* Hypertension poorly controlled on treatment (defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
* Subject with other malignant tumors within 5 years before the screening period, except for cervical carcinoma in situ, breast carcinoma in situ and cutaneous basal cell carcinoma that have received appropriate treatment and met the recovery criteria;
* Subject with a history of autoimmune diseases [such as, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (hypothyroidism without clinical symptoms or hypothyroidism caused by chemoradiotherapy can be included), subjects with vitiligo or recovered asthma can be included without any intervention, and subjects with asthma requiring bronchodilators for medical intervention cannot be included];
* Subject who has previously received similar therapeutic tumor vaccines;
* Subject with congenital or acquired immunodeficiency;
* Subject still participating in other clinical trials and not enrolled at the screening period;
* Subject who is unable or unwilling to comply with the study protocol due to potential health, mental or social conditions in the opinion of the investigator;
* Other conditions that, in the opinion of the investigator, would make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MTD or Clinical recommended dose | Baseline through 90 days after last XH001 dose, up to 6 months
DLT | Cycle 1, up to 21 days
  Rate of Dose Limiting Toxicities
Incidence and degree of Adverse Events and Serious Adverse Events [Safety] | Baseline through 90 days after last sintilimab dose, up to 1 year
  Incidence and degree of participants with adverse events(CTCAE 5.0)

SECONDARY OUTCOMES:
Antigen-Specific T-cell Responses in Peripheral Blood | Baseline through last sintilimab dose, up to 1 year
Number of specific immune response T cells | Baseline through last sintilimab dose, up to 1 year
  Pharmacodynamics parameter
Overall Response Rate (ORR) | up to 2 years
Best Overall Response (BOR) | up to 2 years
Disease Control Rate (DCR) | up to 2 years
Progression Free Survival (PFS) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianming XU, Dr., Principal Investigator — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No